CLINICAL TRIAL: NCT03816449
Title: Influence of Specifically Designed Exercise Program on Serum Matrix Metalloproteinases and Functional Status in Women With Postmenopausal Osteoporosis
Brief Title: Influence of Exercise Program on Serum Matrix Metalloproteinases and Functional Status in Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Responsible Party: Principal Investigator, Tamara Filipovic, Assistant of physical and rehabilitation medicine, Principal investigator, Institut za Rehabilitaciju Sokobanjska Beograd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: : IRehabilitaciju
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Influence of Specifically Designed Exercise Program on Serum Matrix Metalloproteinases and Functional Status in Women With Postmenopausal Osteoporosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): Experimental group will include postmenopausal women who will practice following exercise program:aerobic exercise, resistance training and balance exercise. Aerobic exercise will be conducted as a dose walk, 3-5 km / h, approximately 70% of maximal heart rate, about 50 minutes per day, five days per week, for 12 weeks. Resistance training and balance exercises will be conducted as a group program and will involve exercises to strengthen the muscles of the upper and lower extremities and balance exercises. The intensity of the training will be increased weekly, starting from 3-5 repeating load and its own weight, up to 8-12 repetitions with straps. Frequency of training will be 3 times per week, will last 70 minutes per day, for 12 weeks.
  Interventions: Other: exercises
- control group (Placebo Comparator): Control group will include about postmenopausal women who will not practice exercise program (aerobic exercise, resistance training and balance exercise) .They will continue to carry out activities of daily living, which are conducted daily before inclusion in the study. These patients will be asked to not include in any other program of physical activity and exercise during the research period (12 weeks). After this period, patients will be offered to participate in the same exercise program that had patients from the experimental group.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Aerobic exercise will be conducted as a dose walk, 3-5 km / h, lasting 50 minutes per day, least five days per week, for 12 weeks. The intensity of the training will be around 70% of the maximal heart rate.
  Resistance training and balance exercises will be conducted as a group program and will involve exercises to strengthen the muscles of the upper and lower extremities and balance exercises. The intensity of the training will be increased on weekly, starting from 3-5 repeating load and its own weight, up to 8-12 repetitions and load straps. Progression and maintenance load tapes will be carried out depending on the capacity of individualized persons. Frequency of training will be 3 times a week,will last 70 minutes per day for 12 weeks.

SUMMARY:
Osteoporosis is a chronic, systemic and the most frequently metabolic bone disease, characterized by low bone mass and microarchitectural remodeling of bone, which results in a greater fragility of the bone and risk of fracture. With the purpose of explaining the patophysiological mechanisms responsible for osteoporosis, it is necessary to determine the factors that influence on the activity and differentiation of osteoblasts and osteoclasts, as well as their dynamic change depending on the use of an appropriate treatment.

According to the recommendations of the International Association for osteoporosis (the National Osteoporosis Fondation- NOF) the treatment of osteoporosis includes pharmacological and non-pharmacological treatment of. Pharmacological includes a range of different drug, where the bisphosphonates, non-hormonal antiresorptive drugs, present gold standard in the treatment of postmenopausal osteoporosis . Non-pharmacological treatment implies the daily physical activity and the specific exercise program, for the purpose of slowing or stopping the loss of bone mass, improve balance, and reduce the risk of falling and fractures.

It is known that the mechanical loading of the bone has to be strong enough to achieve the effect of osteogenesis. The load due to the long bones of gravity and the tension force produced by the muscular activity, are the natural stimulus for maintenance of bone mass and muscle strength. This can be achieved by practice involving the activities in which the net mass of the body constitutes an additional load (so-called. "Weight-bearing exercises"), as well as exercise resistance from.

Exercise with one's own mass include actions to counter gravity in an upright standing position, and then may be a stronger (high-impact) collides with the substrate (e.g., jumping) and the lower (low-impact) collides with the substrate (e.g., walking). Aerobic exercise, especially walking, is the most common type of intervention because of the ease administration and safety.

Resistance training is another effective type of exercises that can affect the maintenance or improvement of bone mineral density, with the most frequently applied with the combination of the dynamic resistance exercises that engage multiple joints, large groups of muscles, and the burden on the hips and the spine. In order to strength training, with the aim of maintaining and stimulating bone mineral density had the best effect, it is necessary to include the basic principles of specificity, load and progression. Training should be directed to the adaptation of a specific part of the body, should be sufficiently intense to and beyond the common load, and a variety of progressive enough. Progression loads should be slow and gradual to avoid injury. We assumed that this type of exercise can be achieved by changing the activity of serum matrix metalloproteinases.

It has been proven that in the process of remodeling of the extracellular matrix of the bone, matrix-metalloproteinases play an important role, both, the occurrence of bone as well as in pathological processes of bone resorption . Also, it is known that metalloproteinases, particularly the MMP-2 and MMP-9 play a significant role in the development of skeletal muscle recovery from injury or remodeling of the same after exercise.Taking into account the results of the latest studies on the role of metalloproteinases in the development and remodeling of bone, also and muscle, we assumed that the value of metalloproteinases could serve as markers for early assessment of treatment response of patients with osteoporosis. In our study, we will follow the changes of serum levels of metalloproteinases as well as tissue inhibitor of matrix metalloproteinases 1 (TIMP-1) in the serum of patients with postmenopausal osteoporosis, which have prescribed bisphosphonates, before and after application to the specifically designed exercise program . A functional genetic polymorphisms (PM), by modulating the expression of the MMP can be associated with a differential response to the application of our patients of the same exercise program. Specifically designed exercise program in patients with osteoporosis, which affects the increase in BMD and muscle strength, can be associated with a specific MMP genotyp . In our research we will follow the influence of polymorphisms of the mentioned metalloproteinases on the efficacy of the treatment (the specifically designed exercise program ) in patients with postmenopausal osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a chronic, systemic and the most frequently metabolic bone disease, characterized by low bone mass and microarchitectural remodeling of bone, which results in a greater fragility of the bone and risk of fracture. With the purpose of explaining the patophysiological mechanisms responsible for osteoporosis, it is necessary to determine the factors that influence on the activity and differentiation of osteoblasts and osteoclasts, as well as their dynamic change depending on the use of an appropriate treatment.

According to the recommendations of the International Association for osteoporosis (the National Osteoporosis Fondation- NOF) the treatment of osteoporosis includes pharmacological and non-pharmacological treatment of. Pharmacological includes a range of different drug, where the bisphosphonates, non-hormonal antiresorptive drugs, present gold standard in the treatment of postmenopausal osteoporosis . Non-pharmacological treatment implies the daily physical activity and the specific exercise program, for the purpose of slowing or stopping the loss of bone mass, improve balance, and reduce the risk of falling and fractures.

It is known that the mechanical loading of the bone has to be strong enough to achieve the effect of osteogenesis. The load due to the long bones of gravity and the tension force produced by the muscular activity, are the natural stimulus for maintenance of bone mass and muscle strength. This can be achieved by practice involving the activities in which the net mass of the body constitutes an additional load (so-called. "Weight-bearing exercises"), as well as exercise resistance from.

Exercise with one's own mass include actions to counter gravity in an upright standing position, and then may be a stronger (high-impact) collides with the substrate (e.g., jumping) and the lower (low-impact) collides with the substrate (e.g., walking). Aerobic exercise, especially walking, is the most common type of intervention because of the ease administration and safety.

Resistance training is another effective type of exercises that can affect the maintenance or improvement of bone mineral density, with the most frequently applied with the combination of the dynamic resistance exercises that engage multiple joints, large groups of muscles, and the burden on the hips and the spine. In order to strength training, with the aim of maintaining and stimulating bone mineral density had the best effect, it is necessary to include the basic principles of specificity, load and progression. Training should be directed to the adaptation of a specific part of the body, should be sufficiently intense to and beyond the common load, and a variety of progressive enough. Progression loads should be slow and gradual to avoid injury. We assumed that this type of exercise can be achieved by changing the activity of serum matrix metalloproteinases.

It has been proven that in the process of remodeling of the extracellular matrix of the bone, matrix-metalloproteinases play an important role, both, the occurrence of bone as well as in pathological processes of bone resorption . Also, it is known that metalloproteinases, particularly the MMP-2 and MMP-9 play a significant role in the development of skeletal muscle recovery from injury or remodeling of the same after exercise.Taking into account the results of the latest studies on the role of metalloproteinases in the development and remodeling of bone, also and muscle, we assumed that the value of metalloproteinases could serve as markers for early assessment of treatment response of patients with osteoporosis. In our study, we will follow the changes of serum levels of metalloproteinases as well as tissue inhibitor of matrix metalloproteinases 1 (TIMP-1) in the serum of patients with postmenopausal osteoporosis, which have prescribed bisphosphonates, before and after application to the specifically designed exercise program . A functional genetic polymorphisms (PM), by modulating the expression of the MMP can be associated with a differential response to the application of our patients of the same exercise program. Specifically designed exercise program in patients with osteoporosis, which affects the increase in BMD and muscle strength, can be associated with a specific MMP genotyp . In our research we will follow the influence of polymorphisms of the mentioned metalloproteinases on the efficacy of the treatment (the specifically designed exercise program ) in patients with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis, diagnosed by central osteodensitometry in patients aged between 65 and 70 years, and osteoporosis diagnosed by central osteodensitometry in patients aged less than 65 under the risk factors for osteoporosis (early menopause, late menopause, extended amenorrhea, a positive family history related to energy fracture, etc., as defined by the NOF)

Exclusion Criteria:

* Perimenopausal status (with the appearance of irregular cycles in the past year), metabolic bone disease, which can be a cause of secondary osteoporosis, hyperparathyroidism, verified oncological diseases, the use of corticosteroids for more than 3 months, hormonal therapy, hepatic dysfunction and kidney, heart and signs of respiratory insufficiency, participation in any exercise program in the last 2 months, including the rapid motion of 3km / h at least 3 times a week.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in enzyme activity of matrix metalloproteinase-2 , matrix metalloproteinase- 9 and tissue inhibitor of matrix metalloproteinase 1 (TIMP-1) in serum | Change measures ( "baseline , 4 weeks and 12 weeks")
  For the following biochemical parameters, patients will be taken peripheral blood (on an empty stomach), centrifuged at 3000 rpm / min, split up into aliquots (serum and plasma) and kept in the freezer (at -20 ° C) for determination the following parameters.
Functional assessment of the musculoskeletal system using Timed-Up and Go Test" (TUG test) | Change measures ( "baseline , 4 weeks and 12 weeks")
  "Timed-Up and Go Test" is an effective method for estimating the motion and function of the musculoskeletal system, in patients with osteoporosis. Performed by being the person required to get up from the chair usual height with backrest (seat height about 46 cm, height of armrest 65 cm) to walk 3 m normal walking speed, turned back to the chair and then sit on the same. Typically this activity is carried out in less than 12 seconds, over this is considered to be an increased risk for the drop and reduced muscle function.
Functional assessment of the musculoskeletal system using "Chair Rising Test ". | Change measures ( "baseline , 4 weeks and 12 weeks")
  "Chair Rising Test "is a simple test that is used to assess the strength of the lower extremities and is often used for assessing the risk of falls in patients with osteoporosis. It is performed by the request from the person to get up from the chair height and common to sit on the same 5 times as fast as possible, without using hands. His hands were clasped in front of her chest. Inability to 5 times stand up or sit down, or over the test duration of 10 seconds is interpreted as a decrease in muscular strength and increased risk of falling.
Functional assessment of the musculoskeletal system using "One-Leg Stance Test". | Change measures ( "baseline , 4 weeks and 12 weeks")
  One-Leg Stance Test" (OLST) is a clinical tool that is used for a quantitative assessment of static balance, and consequently the risk assessment for the pad and the functional dependence. Is performed so that the respondent is required to stand on one foot (dominant) to a stable platform without the support and aids, with eyes open, and the hands to the body, wherein a stop watch measuring time for which the respondent can perform a task in seconds. It will be made of two measurements, wherein the best value is adopted in the assay and assessment of the risk is determined according to the set values for a given age.

SECONDARY OUTCOMES:
Detection of genotypes for the polymorphisms: rs243866 in the gene for MMP-2 | Change measures ( "baseline and 12 weeks")
  Detection of genotypes for the polymorphisms: rs243866 in the gene for MMP-2 will be effected Real time PCR method with the use of standardized TaqMan®SNP Genotyping assay.
Detection of genotypes of rs3918242 polymorphism in the MMP-9 | Change measures ( "baseline and 12 weeks")
  The genotypes of rs3918242 polymorphism in the MMP-9 gene will be determined by reaction of the polymerization chain (PCR) and restriction products of the reaction the restriction enzyme. Analysis of the genotypes will be performed after electrophoretic separation in 8% polyacrylamide gels nondenaturated, coloring Sybr®safe DNA stain and illumination under UV transillumination.

CONTACTS AND LOCATIONS:
Locations (1):
- Tamara Filipovic, Belgrade, Serbia

REFERENCES:
- [Derived] Filipovic T, Gopcevic K, Dimitrijevic S, Hrkovic M, Backovic A, Lazovic M. Effects of 12-Week Exercise Program on Enzyme Activity of Serum Matrix Metalloproteinase-9 and Tissue Inhibitor of Metalloproteinase-1 in Female Patients with Postmenopausal Osteoporosis: A Randomized Control Study. Biomed Res Int. 2020 Jan 30;2020:9758289. doi: 10.1155/2020/9758289. eCollection 2020. PMID 32071923